CLINICAL TRIAL: NCT01115803
Title: A Phase 1b Trial of LY2584702 in Combination With Erlotinib or Everolimus in Patients With Solid Tumors
Brief Title: A Study of LY2584702 With Erlotinib or Everolimus in Participants With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Primary objective has been met; safety and pharmacokinetics have been characterized.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 12531; I3G-MC-JGCB (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-04-22; First posted 2010-05-04 (Estimated); Results first posted 2019-01-18 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Metastases, Neoplasm; Carcinoma, Non-small Cell Lung; Renal Cell Carcinoma; Neuroendocrine Tumors
Keywords: Advanced Cancer; Metastatic Cancer; Non-Small Cell Lung Cancer; Renal Cell Carcinoma; Neuroendocrine Tumors
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Neuroendocrine Tumors | interventions — LY2584702; Erlotinib Hydrochloride; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: LY2584702 + Erlotinib (Experimental): Participants received 50 mg LY2584702 once daily (QD )+ 150 mg Erlotinib QD, 50 mg LY2584702 twice daily (BID) + 150 mg Erlotinib QD, 100 mg LY2584702 BID + 150 mg Erlotinib QD and 75 mg LY2584702 BID + 150 mg Erlotinib QD.
  Interventions: Drug: LY2584702; Drug: Erlotinib
- Arm B: LY2584702 + Everolimus (Experimental): Participants received 50 mg LY2584702 QD + 10 mg Everolimus QD, 100 mg LY2584702 QD + 10 mg Everolimus QD and 50 mg LY2584702 BID + 10 mg Everolimus QD.
  Interventions: Drug: LY2584702; Drug: Everolimus

INTERVENTIONS:
Drug: LY2584702 — Supplied as 25 milligrams (mg) and 100 mg capsules, administered orally for two 28-day cycles.
Drug: Erlotinib — Supplied as 25 mg, 100 mg, or 150 mg tablets, administered orally, daily for two 28-day cycles.
  Starting dose is 150mg. Doses may be decreased in 50mg increments if necessary due to toxicity.
  Arms: Arm A: LY2584702 + Erlotinib
Drug: Everolimus — Supplied as 5 mg or 10 mg tablets, administered orally, daily for two 28-day cycles.
  Arms: Arm B: LY2584702 + Everolimus

SUMMARY:
Study I3G-MC-JGCB (JGCB) is a multicenter, nonrandomized, open-label, dose-escalation Phase 1b study of LY2584702 in combination with either erlotinib or everolimus.

DETAILED DESCRIPTION:
Study JGCB will consist of the following parts:

Part 1 - Dose Escalation to maximum tolerated dose in each arm.

Arm A - LY2584702 + Erlotinib in participants with advanced or metastatic cancer.

Arm B - LY2584702 + Everolimus in participants with advanced or metastatic cancer.

Part 2 - Dose Confirmation of maximum tolerated dose from each arm in Part 1.

Arm A - LY2584702 + Erlotinib in participants with advanced or metastatic non-small cell lung cancer.

Arm B - LY2584702 + Everolimus in participants with advanced renal cell carcinoma after treatment failure with sunitinib or sorafenib, or advanced neuroendocrine tumors.

ELIGIBILITY:
Inclusion Criteria:

* Dose Escalation portion (Part 1): have histological or cytological evidence of a diagnosis of cancer that is advanced and/or metastatic disease (including Non-Hodgkin's Lymphoma) for which no proven effective therapy exists.
* Dose Confirmation portion (Part 2): have histological or cytological evidence of:

  1. Arm A: advanced or metastatic non-small cell lung cancer after failure of at least one prior chemotherapy regimen.
  2. Arm B: advanced renal cell carcinoma after failure of treatment with sunitinib or sorafenib, or advanced neuroendocrine tumors.
* Have the presence of measurable or nonmeasurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) or the Revised Response Criteria for Malignant Lymphoma.

  1. Dose Escalation portion (Part 1): participants may have measurable or nonmeasurable disease.
  2. Dose Confirmation portion (Part 2): participants must have measurable disease.
* Have adequate organ function including:

  1. Hematologic: absolute neutrophil count (ANC) greater than or equal to 1.5 x 10⁹/liters (L), platelets greater than or equal to 100 x 10⁹/L, and hemoglobin greater than or equal to 8 grams/deciliter (g/dL).
  2. Hepatic: bilirubin less than or equal to 1.5 times upper limits of normal (ULN); alanine transaminase (ALT) and aspartate transaminase (AST) less than or equal to 2.5 times ULN. If the liver has tumor involvement, AST and ALT equaling less than or equal to 5 times ULN are acceptable. Participants with bone metastases may enter with alkaline phosphatase values less than or equal to 5 times ULN, as long as other hepatic parameters meet inclusion criteria.
  3. Renal: Serum creatinine less than or equal to 1.5 times ULN or calculated creatinine clearance >45 milliliter/minute (ml/mn).
* Have a performance status of less than or equal to 1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, cancer-related hormonal therapy, or other investigational therapy for at least 2 weeks (3 weeks for myelosuppressive agents) prior to study enrollment, and have recovered from the acute effects of therapy. At the discretion of the investigator, participants with prostate cancers progressing under luteinizing hormone-releasing hormone (LHRH) agonists therapy, and participants with adrenal carcinomas using mitotane, may have that treatment continued while receiving study drug.

Exclusion Criteria:

* Have received treatment with a drug that has not received regulatory approval for any indication within 14 or 21 days of the initial dose of study drug for a nonmyelosuppressive or myelosuppressive agent, respectively.
* Have serious preexisting medical conditions that, in the opinion of the investigator, would preclude participation in this study.
* Have symptomatic central nervous system (CNS) malignancy or metastasis. Participants with treated CNS metastases are eligible provided their disease is radiographically stable and asymptomatic, and they are not currently receiving corticosteroids and/or anticonvulsants. Screening of asymptomatic participants without history of CNS metastasis is not required.
* Concomitant treatment by strong cytochrome P450 (CYP) 3A4 inhibitors or CYP3A4 inducers.
* Have an acute or chronic leukemia.
* Have received an autologous or allogeneic stem-cell transplant within 75 days of the initial dose of study drug. In addition, recipients of an allogeneic stem-cell transplant must have discontinued immunosuppressive therapy at least 24 hours before study drug administration with no more than Grade 1 acute graft-versus-host disease.
* For Dose Confirmation portion (Part 2): have previously received erlotinib for Arm A or everolimus for Arm B.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois, United States
- France (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bordeaux
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Villejuif

REFERENCES:
- [Derived] Hollebecque A, Houede N, Cohen EE, Massard C, Italiano A, Westwood P, Bumgardner W, Miller J, Brail LH, Benhadji KA, Soria JC. A phase Ib trial of LY2584702 tosylate, a p70 S6 inhibitor, in combination with erlotinib or everolimus in patients with solid tumours. Eur J Cancer. 2014 Mar;50(5):876-84. doi: 10.1016/j.ejca.2013.12.006. Epub 2014 Jan 20. PMID 24456794

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A 2 phase study, a dose escalation phase and a dose confirmation phase. The dose confirmation phase was not initiated. Participant flow reports those participants who discontinued from study drug. Participants who completed 1 cycle of treatment, had the required assessment or an adverse event (AE) were considered to have completed the study.
Groups:
- Arm A - 50 mg LY2584702 QD + 150 mg Erlotinib QD: 50 milligrams (mg) LY2584702 administered orally once daily (QD) plus 150 mg erlotinib administered orally QD for two 28-day cycles.
- Arm A - 50 mg LY2584702 BID + 150 mg Erlotinib QD: 50 mg LY2584702 administered orally twice daily (BID) plus 150 mg erlotinib administered orally QD for two 28-day cycles.
- Arm A - 100 mg LY2584702 BID + 150 mg Erlotinib QD: 100 mg LY2584702 administered orally BID plus 150 mg erlotinib administered orally QD for two 28-day cycles.
- Arm A - 75 mg LY2584702 BID + 150 mg Erlotinib QD: 75 mg LY2584702 administered orally BID plus 150 mg erlotinib administered orally QD for two 28-day cycles.
- Arm B - 50 mg LY2584702 QD + 10 mg Everolimus QD: 50 mg LY2584702 administered orally QD plus 10 mg everolimus administered orally QD for two 28-day cycles.
- Arm B - 100 mg LY2584702 QD + 10 mg Everolimus QD: 100 mg LY2584702 administered orally QD plus 10 mg everolimus administered orally QD for two 28-day cycles.
- Arm B - 50 mg LY2584702 BID + 10 mg Everolimus QD: 50 mg LY2584702 administered orally BID plus 10 mg everolimus administered orally QD for two 28-day cycles.
Period: Overall Study
Arm/Group | Arm A - 50 mg LY2584702 QD + 150 mg Erlotinib QD | Arm A - 50 mg LY2584702 BID + 150 mg Erlotinib QD | Arm A - 100 mg LY2584702 BID + 150 mg Erlotinib QD | Arm A - 75 mg LY2584702 BID + 150 mg Erlotinib QD | Arm B - 50 mg LY2584702 QD + 10 mg Everolimus QD | Arm B - 100 mg LY2584702 QD + 10 mg Everolimus QD | Arm B - 50 mg LY2584702 BID + 10 mg Everolimus QD
Started | 4 | 5 | 3 | 5 | 3 | 3 | 6
Received at Least 1 Dose of Study Drug | 4 | 5 | 3 | 5 | 3 | 3 | 6
Completed | 4 | 5 | 2 | 5 | 3 | 3 | 4
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive Disease during Cycle1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - 50 mg LY2584702 QD + 150 mg Erlotinib QD | Arm A - 50 mg LY2584702 BID + 150 mg Erlotinib QD | Arm A - 100 mg LY2584702 BID + 150 mg Erlotinib QD | Arm A - 75 mg LY2584702 BID + 150 mg Erlotinib QD | Arm B - 50 mg LY2584702 QD + 10 mg Everolimus QD | Arm B - 100 mg LY2584702 QD + 10 mg Everolimus QD | Arm B - 50 mg LY2584702 BID + 10 mg Everolimus QD | Total
Number analyzed (Participants) | 4 | 5 | 3 | 5 | 3 | 3 | 6 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (7.97) | 61.4 (7.86) | 52.3 (11.02) | 63.0 (3.39) | 49.0 (7.55) | 47.7 (16.01) | 47.5 (16.17) | 54.0 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 1 | 2 | 2 | 3 | 15
  Male | 1 | 3 | 1 | 4 | 1 | 1 | 3 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 3 | 5 | 3 | 3 | 5 | 26
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 4 | 3 | 3 | 5 | 2 | 3 | 4 | 24
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 4
  France | 4 | 4 | 2 | 5 | 3 | 3 | 4 | 25

OUTCOME MEASURES:

1. Primary Outcome: Recommended Dose for Phase 2 Studies
Description: The recommended dose for the Phase 2 (Dose Confirmation Phase) study was determined by safety assessment. Doses were escalated following the assessment for toxicity based on Common Terminology Criteria for Adverse Events (CTCAE v4.0). Any adverse events (AE) that were possibly related to LY2584702 were considered toxicities. The Phase 2 dose of LY2584702 was not determined due to unacceptable toxicities of LY2584702 in combination with erlotinib or everolimus in Phase 1 of the study.
Time Frame: Baseline up to 6 cycles of 28 days
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: milligrams (mg)
Groups:
- LY2584702 + Erlotinib: Escalating doses of LY2584702 began with 50 milligrams (mg) and increased up to 200 mg total daily dose were administered orally in combination with erlotinib.
- LY2584702+Everolimus: Escalating doses of LY2584702 began with 50 mg and increased up to 100 mg total daily dose were administered orally in combination with everolimus.
Arm/Group | LY2584702 + Erlotinib | LY2584702+Everolimus
Number analyzed (Participants) | 17 | 12
milligrams (mg) | NA — The Phase 2 dose of LY2584702 in combination with erlotinib was not determined. | NA — The Phase 2 dose of LY2584702 in combination with everolimus was not determined.

2. Secondary Outcome: Clinically Significant Effects (Number of Participants With Adverse Events)
Description: Clinically significant events were defined as serious adverse events (SAEs) and other non-SAEs regardless of causality. A summary of serious and other non SAEs regardless of causality is located in the Reported Adverse Event module.
Time Frame: Baseline up to 7 months
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - 50 mg LY2584702 QD + 150 mg Erlotinib QD | Arm A - 50 mg LY2584702 BID + 150 mg Erlotinib QD | Arm A - 100 mg LY2584702 BID + 150 mg Erlotinib QD | Arm A - 75 mg LY2584702 BID + 150 mg Erlotinib QD | Arm B - 50 mg LY2584702 QD + 10 mg Everolimus QD | Arm B - 100 mg LY2584702 QD + 10 mg Everolimus QD | Arm B - 50 mg LY2584702 BID + 10 mg Everolimus QD
Number analyzed (Participants) | 4 | 5 | 3 | 5 | 3 | 3 | 6
Participants
  SAEs | 1 | 2 | 2 | 3 | 2 | 2 | 2
  Non-SAEs | 4 | 5 | 3 | 5 | 3 | 3 | 6

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the date of enrollment to the date of objectively determined progressive disease (PD) or death whichever comes first. Censoring of PFS was defined as participants not known to have died as of the data cut-off date and who did not have objective PD, PFS was censored at the date of the last objective assessment; for participants who received subsequent systematic anticancer therapy (after discontinuation from study treatment) prior to objectively determined disease progression, PFS was censored at the date of the last objective progression-free disease assessment prior to post discontinuation of therapy. PFS was not analyzed due to different tumor types and different doses.
Time Frame: Baseline to disease progression or death or up to 166 days postbaseline
Population: Zero participants were analyzed as no data collected.
Arm/Group | Arm A - 50 mg LY2584702 QD + 150 mg Erlotinib QD | Arm A - 50 mg LY2584702 BID + 150 mg Erlotinib QD | Arm A - 100 mg LY2584702 BID + 150 mg Erlotinib QD | Arm A - 75 mg LY2584702 BID + 150 mg Erlotinib QD | Arm B - 50 mg LY2584702 QD + 10 mg Everolimus QD | Arm B - 100 mg LY2584702 QD + 10 mg Everolimus QD | Arm B - 50 mg LY2584702 BID + 10 mg Everolimus QD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR) [Response Rate (RR)]
Description: Response was determined using Response Evaluation Criteria In Solid Tumors (RECIST v1.1) criteria. CR was defined as the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeters (mm) and normalization of tumor marker level of non-target lesions; PR was defined as at least a 30% decrease in sum of longest diameter of target lesions.
Time Frame: Baseline to disease progression or death or up to 6 cycles of 28 days
Population: All participants who received at least 1 dose of study drug and assessed for RR.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Arm A - 50 mg LY2584702 QD + 150 mg Erlotinib QD: 50 milligram (mg) LY2584702 administered orally once daily (QD) plus 150 mg erlotinib administered orally QD for two 2 28-day cycles.
- Arm A - 50 mg LY2584702 (BID) + 150 mg Erlotinib QD: 50 mg LY2584702 administered orally twice daily (BID) plus 150 mg erlotinib administered orally QD for two 28-day cycles.
Arm/Group | Arm A - 50 mg LY2584702 QD + 150 mg Erlotinib QD | Arm A - 50 mg LY2584702 (BID) + 150 mg Erlotinib QD | Arm A - 100 mg LY2584702 BID + 150 mg Erlotinib QD | Arm A - 75 mg LY2584702 BID + 150 mg Erlotinib QD | Arm B - 50 mg LY2584702 QD + 10 mg Everolimus QD | Arm B - 100 mg LY2584702 QD + 10 mg Everolimus QD | Arm B - 50 mg LY2584702 BID + 10 mg Everolimus QD
Number analyzed (Participants) | 4 | 5 | 2 | 3 | 3 | 3 | 3
percentage of participants | 0 [NA to NA] — No participants achieved PR or CR; confidence interval could not be determined. | 0 [NA to NA] — No participants achieved PR or CR; confidence interval could not be determined. | 0 [NA to NA] — No participants achieved PR or CR; confidence interval could not be determined. | 0 [NA to NA] — No participants achieved PR or CR; confidence interval could not be determined. | 0 [NA to NA] — No participants achieved PR or CR; confidence interval could not be determined. | 0 [NA to NA] — No participants achieved PR or CR; confidence interval could not be determined. | 0 [NA to NA] — No participants achieved PR or CR; confidence interval could not be determined.

5. Secondary Outcome: Pharmacokinetics, Maximum Observed Plasma Concentration (Cmax) of LY2584702
Time Frame: Cycle 1 Day 1 (C1 D1): predose, 0.5, 1, 2, 3, 5, 8 hours postdose and Cycle 1 Day 8 (C1 D8): predose, 0.5, 1, 2, 3, 5, and 8 hours postdose of 28-day cycle
Population: All participants who received at least 1 dose of study drug and had Cmax values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Arm A - 50 mg LY2584702 QD + 150 mg Erlotinib QD: 50 milligram (mg) LY2584702 administered orally once daily (QD) plus 150 mg erlotinib administered orally QD for two 28-day cycles.
Arm/Group | Arm A - 50 mg LY2584702 QD + 150 mg Erlotinib QD | Arm A - 50 mg LY2584702 BID + 150 mg Erlotinib QD | Arm A - 100 mg LY2584702 BID + 150 mg Erlotinib QD | Arm A - 75 mg LY2584702 BID + 150 mg Erlotinib QD | Arm B - 50 mg LY2584702 QD + 10 mg Everolimus QD | Arm B - 100 mg LY2584702 QD + 10 mg Everolimus QD | Arm B - 50 mg LY2584702 BID + 10 mg Everolimus QD
Number analyzed (Participants) | 4 | 4 | 3 | 5 | 3 | 3 | 6
nanograms per milliliter (ng/mL)
  C1 D1, single dose: number analyzed (Participants) | 3 | 4 | 3 | 5 | 3 | 2 | 3
  C1 D1, single dose | 918.24 (42.9) | 999.54 (68.3) | 2421.64 (35.1) | 1768.59 (50.3) | 1192.46 (31.5) | 2286.22 (7.3) | 1569.24 (28.6)
  C1 D8, steady state: number analyzed (Participants) | 4 | 4 | 3 | 4 | 3 | 3 | 6
  C1 D8, steady state | 1125.46 (64.6) | 1636.71 (52.6) | 2709.61 (50.7) | 1967.04 (24.8) | 1169.95 (25.2) | 2260.71 (34.8) | 2109.62 (44.1)

6. Secondary Outcome: Pharmacokinetics, Area Under the Concentration Time Curve (AUC)
Description: AUC from time 0 to 8 hours (AUC0-8) and AUC from time 0 to infinity (AUC0-∞).
Time Frame: Cycle 1 Days 1 (C1 D1) and Cycle 1 Day 8 (C1 D8) of 28-day cycle
Population: All participants who received at least 1 dose of study drug and had AUC values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Arm/Group | Arm A - 50 mg LY2584702 QD + 150 mg Erlotinib QD | Arm A - 50 mg LY2584702 BID + 150 mg Erlotinib QD | Arm A - 100 mg LY2584702 BID + 150 mg Erlotinib QD | Arm A - 75 mg LY2584702 BID + 150 mg Erlotinib QD | Arm B - 50 mg LY2584702 QD + 10 mg Everolimus QD | Arm B - 100 mg LY2584702 QD + 10 mg Everolimus QD | Arm B - 50 mg LY2584702 BID + 10 mg Everolimus QD
Number analyzed (Participants) | 4 | 4 | 3 | 5 | 3 | 3 | 6
nanograms*hours per milliliter (ng*h/mL)
  AUC0-8, D1, single dose: number analyzed (Participants) | 3 | 4 | 3 | 5 | 3 | 2 | 3
  AUC0-8, D1, single dose | 4436.60 (50.6) | 4308.98 (79.8) | 8610.54 (49.4) | 8091.93 (47.8) | 5699.856 (31.9) | 11410.18 (3.9) | 6097.44 (15.9)
  AUC0-8, D8, steady state: number analyzed (Participants) | 4 | 3 | 3 | 4 | 3 | 3 | 6
  AUC0-8, D8, steady state | 5395.96 (70.7) | 7948.43 (50.4) | 15225.08 (43.0) | 13959.74 (45.6) | 5460.80 (23.3) | 11327.33 (34.7) | 10527.68 (44.1)
  AUC0-∞, D1, single dose: number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 2 | 3
  AUC0-∞, D1, single dose | 8699.54 (38.0) | 7627.50 (37.9) | 20813.83 (25.0) | 16254.07 (20.3) | 11386.03 (34.8) | 22343.07 (NA) — Only 2 participants analyzed | 8764.13 (14.1)

7. Secondary Outcome: Number of Participants With Complete Response (CR), Partial Response (PR) or Stable Disease (SD) [Best Overall Response (BOR) (CR+PR+SD)]
Description: BOR was determined using Response Evaluation Criteria In Solid Tumors (RECIST v1.1) criteria. CR was defined as the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeters (mm) and normalization of tumor marker level of non-target lesions; PR was defined as at least a 30% decrease in sum of longest diameter (LD) of target lesions; Progressive Disease (PD) was defined as at least 20% increase in sum of LD of target lesions and minimum 5 mm increase over nadir. SD was defined as small changes that did not meet above criteria.
Time Frame: Baseline up to 112 Days
Population: All participants who received at least 1 dose of study drug and assessed for BOR.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - 50 mg LY2584702 QD + 150 mg Erlotinib QD | Arm A - 50 mg LY2584702 BID + 150 mg Erlotinib QD | Arm A - 100 mg LY2584702 BID + 150 mg Erlotinib QD | Arm A - 75 mg LY2584702 BID + 150 mg Erlotinib QD | Arm B - 50 mg LY2584702 QD + 10 mg Everolimus QD | Arm B - 100 mg LY2584702 QD + 10 mg Everolimus QD | Arm B - 50 mg LY2584702 BID + 10 mg Everolimus QD
Number analyzed (Participants) | 4 | 5 | 2 | 3 | 3 | 3 | 3
Participants | 1 | 1 | 1 | 1 | 0 | 2 | 2

8. Other Pre Specified Outcome: Number of Participants Who Died Due to Progressive Disease Within 30 Days of Study Drug Discontinuation
Time Frame: Within 30 days of study drug discontinuation
Population: Participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - 50 mg LY2584702 QD + 150 mg Erlotinib QD | Arm A - 50 mg LY2584702 BID + 150 mg Erlotinib QD | Arm A - 100 mg LY2584702 BID + 150 mg Erlotinib QD | Arm A - 75 mg LY2584702 BID + 150 mg Erlotinib QD | Arm B - 50 mg LY2584702 QD + 10 mg Everolimus QD | Arm B - 100 mg LY2584702 QD + 10 mg Everolimus QD | Arm B - 50 mg LY2584702 BID + 10 mg Everolimus QD
Number analyzed (Participants) | 4 | 5 | 3 | 5 | 3 | 3 | 6
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Description: Deaths due to progressive disease were not considered to be serious adverse events (SAE) unless the investigator deemed them to be related to the use of the study drug.
Groups:
- Arm A - 50 mg LY2584702 QD + 150 mg Erlotinib QD: 50 milligram (mg) LY2584702 administered orally once daily (QD) plus 150 mg erlotinib administered orally QD for 2 28-day cycles.
- Arm A - 50 mg LY2584702 BID + 150 mg Erlotinib QD: 50 mg LY2584702 administered orally twice daily BID plus 150 mg erlotinib administered orally QD for 2 28-day cycles.
- Arm A - 100 mg LY2584702 BID + 150 mg Erlotinib QD: 100 mg LY2584702 administered orally BID plus 150 mg erlotinib administered orally QD for 2 28-day cycles.
- Arm A - 75 mg LY2584702 BID + 150 mg Erlotinib QD: 75 mg LY2584702 administered orally BID plus 150 mg erlotinib administered orally QD for 2 28-day cycles.
- Arm B - 50 mg LY2584702 QD + 10 mg Everolimus QD: 50 mg LY2584702 administered orally QD plus 150 mg everolimus administered orally QD for 2 28-day cycles.
- Arm B - 100 mg LY2584702 QD + 10 mg Everolimus QD: 100 mg LY2584702 administered orally QD plus 150 mg everolimus administered orally QD for 2 28-day cycles.
- Arm B - 50 mg LY2584702 BID + 10 mg Everolimus QD: 50 mg LY2584702 administered orally BID plus 150 mg everolimus administered orally QD for 2 28-day cycles.
Arm/Group | Arm A - 50 mg LY2584702 QD + 150 mg Erlotinib QD | Arm A - 50 mg LY2584702 BID + 150 mg Erlotinib QD | Arm A - 100 mg LY2584702 BID + 150 mg Erlotinib QD | Arm A - 75 mg LY2584702 BID + 150 mg Erlotinib QD | Arm B - 50 mg LY2584702 QD + 10 mg Everolimus QD | Arm B - 100 mg LY2584702 QD + 10 mg Everolimus QD | Arm B - 50 mg LY2584702 BID + 10 mg Everolimus QD
Serious Adverse Events (participants affected / at risk) | 1/4 | 2/5 | 2/3 | 3/5 | 2/3 | 2/3 | 2/6
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 3/3 | 5/5 | 3/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - 50 mg LY2584702 QD + 150 mg Erlotinib QD (N=4) | Arm A - 50 mg LY2584702 BID + 150 mg Erlotinib QD (N=5) | Arm A - 100 mg LY2584702 BID + 150 mg Erlotinib QD (N=3) | Arm A - 75 mg LY2584702 BID + 150 mg Erlotinib QD (N=5) | Arm B - 50 mg LY2584702 QD + 10 mg Everolimus QD (N=3) | Arm B - 100 mg LY2584702 QD + 10 mg Everolimus QD (N=3) | Arm B - 50 mg LY2584702 BID + 10 mg Everolimus QD (N=6)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Arm A - 50 mg LY2584702 QD + 150 mg Erlotinib QD (N=4) | Arm A - 50 mg LY2584702 BID + 150 mg Erlotinib QD (N=5) | Arm A - 100 mg LY2584702 BID + 150 mg Erlotinib QD (N=3) | Arm A - 75 mg LY2584702 BID + 150 mg Erlotinib QD (N=5) | Arm B - 50 mg LY2584702 QD + 10 mg Everolimus QD (N=3) | Arm B - 100 mg LY2584702 QD + 10 mg Everolimus QD (N=3) | Arm B - 50 mg LY2584702 BID + 10 mg Everolimus QD (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (3) | 4 (6) | 2 (4) | 2 (3) | 3 (4)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (3) | 4 (4) | 2 (2) | 2 (2) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 3 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 2 (4) | 3 (3)
Asthenia (General disorders) | 3 (3) | 3 (3) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 4 (4)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Cytolytic hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0/3 (0) | 0/2 (0) | 0/2 (0) | 1/1 (1) | 0/2 (0) | 0/2 (0) | 0/3 (0)
Vulvovaginitis (Infections and infestations) | 1/3 (1) | 0/2 (0) | 0/2 (0) | 0/1 (0) | 0/2 (0) | 0/2 (0) | 0/3 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coagulation factor v level decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram repolarisation abnormality (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 5 (5) | 2 (2) | 3 (3) | 2 (3) | 0 (0) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Micturition disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study terminated early. Dose confirmation, Part B, was not initiated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days